CLINICAL TRIAL: NCT07007273
Title: Pembrolizumab for Advanced Cutaneous Sarcomas Not Including Angiosarcoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-23318
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Cutaneous Sarcoma
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab Treatment (Experimental): Pembrolizumab 200 mg will be administered as 30-minute IV infusion every 21 days (3 weeks).
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Outpatient infusion
  Other Names: Keytruda

SUMMARY:
This is a single arm, open-label phase II study to assess the efficacy of single agent pembrolizumab for the treatment of advanced cutaneous sarcomas. Adult patients ≥18 years old who have been diagnosed with an advanced cutaneous sarcoma without regard to race, ethnicity, and/or gender. Approximately N=17 patients are planned to be enrolled. Pembrolizumab 200 mg will be administered as 30-minute IV infusion every 21 days (3 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of soft tissue sarcoma, not including angiosarcoma, will be enrolled on study. The primary tumor site must be deemed to be cutaneous or dermal in the opinion of the treating investigator (note the primary tumor site does NOT need to be present at the time of screening, i.e., may have been previously resected but recurred and/or metastasized).
* Participants must have metastatic or advanced disease which could include recurrent, unresectable or multifocal lesions or in which resection would result in unacceptable morbidity per the treating investigator.
* Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Archival tumor tissue sample or newly obtained [core, punch, incisional, or excisional] biopsy of a tumor lesion not previously irradiated is available. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue.
* Prior oncologic therapy is allowable but not required. Must be at least 4 weeks since prior systemic anti-cancer therapy including investigational agents prior to start of study treatment. For prior tyrosine kinase inhibitor therapy, 3 drug half-lives may instead be used for this criterion (if shorter). Must be at least 2 weeks since prior radiotherapy prior to start of study treatment.
* Have an ECOG performance status ≤ 1.
* Participants must have adequate organ and marrow function as defined in the protocol.
* HIV-infected participants must have well-controlled HIV on ART.
* Participants who are HBsAg positive are eligible if they have received HBV anti-viral therapy for at least 4 weeks, and have undetectable HBV viral load prior to randomization.
* Participants with a history of HCV infection are eligible if HCV viral load is undetectable at screening.
* Participants with treated brain metastases are eligible if follow-up brain imaging after central nervous system- (CNS-) directed therapy shows no evidence of progression for at least 4 weeks by repeat imaging, clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study therapy.
* Participants with a prior or concurrent malignancy are eligible for this trial if the malignancy is not progressing and has not required therapy in the past 3 years.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).
* Participants who have not recovered from adverse events (AEs) due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1), with the exception of alopecia or participants who have ≤Grade 2 neuropathy.
* Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of other vaccine types is allowed.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Has active autoimmune disease that has required systemic treatment in the past 2 years except replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid)
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has an active infection requiring systemic therapy.
* Has not adequately recovered from major surgery or has ongoing surgical complications.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Participants with psychiatric illness/social situations that would limit compliance with study requirements.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
* Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 3 years
  Objective response rate will be determined by RECIST 1.1.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 3 years
  Overall survival (OS) will be assessed by Kaplan-Meier method.
Progression Free Survival (PFS) | Up to 3 years
  Progression free survival (PFS) will be assessed by Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Brohl, MD, Principal Investigator — Moffitt Cancer Center
Locations (3):
- United States (3):
  - Moffitt Cancer Center, Tampa, Florida
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided